CLINICAL TRIAL: NCT03830684
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter and Phase Ⅱa Clinical Trial for the Effectiveness and Safety of Baicalein Tablets in the Treatment of Improve Other Aspects of Healthy Adult With Influenza Fever
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HQS201801/PRO
Record Dates: First submitted 2018-12-12; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baicalein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose group (Experimental): Baicalein Tablets group
  Interventions: Drug: Baicalein Tablets 400mg
- high-dose group (Experimental): Baicalein Tablets group
  Interventions: Drug: Baicalein Tablets 600mg
- placebo group (Placebo Comparator): control group
  Interventions: Drug: blank control 0mg

INTERVENTIONS:
Drug: Baicalein Tablets 400mg — 4 Baicalein Tablets and 2 placebo per time, three times a day
  Arms: low-dose group
Drug: Baicalein Tablets 600mg — 6 Baicalein Tablets per time, three times a day
  Arms: high-dose group
Drug: blank control 0mg — 6 placebo per time, three times a day
  Arms: placebo group

SUMMARY:
This study in order to evaluate the Baicalein Tablets' safety and efficiency for audit with influenza

DETAILED DESCRIPTION:
This study in order to evaluate the Baicalein Tablets' safety and efficiency for audit with influenza, The trial designed by randomized, double-blind, placebo-controlled, multicenter and optimal efficiency. Subjects will be randomly assigned to low-dose group, high-dose group or placebo group as 1:1:1 proportionally, planned to enroll 180 subjects, each group enroll 60 subjects. The primary indicator is the time of fever relieving, comparison after the second visit. The secondary indicator are symptom alleviating time of influenza, percentage of subjects with influenza complications, percentage of antipyretic drugs used, percentage of virus positive to negative, comparison at the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meet the diagnostic criteria for influenza（non-severe）; 2.Fever to take medicine for the first time, The patient's maximum temperature (axillary temperature) is over 38℃; 3.The rapid virus antigen test of nasal swab was positive; 4.Course of disease ≤ 24 hours(The definition of course of disease is the time from fever to take investigational product for the first time); 5.Aged 18 to 65 years old(include 18 and 65), all genders; 6.Sign the informed consent form.

Exclusion Criteria:

* 1.The patients with severe influenza or complication (e.g. secondary bacterial pneumonia, pneumonia caused by other pathogens or other viral pneumonia); 2.The patients with other acute upper respiratory tract infection (e.g. acute pharyngitis, tonsillitis, rhinitis and nasosinuitis); 3.Allergic to baicalin and its analogue, Paracetamol tablets, or allergic people; 4.Patients with any of the following risk factors:

  1. Residents living in long-term care facilities (e.g. welfare house, sanatorium);
  2. Combined with chronic respiratory diseases (e.g. bronchial asthma, chronic obstrctive palmonary diseases);
  3. Combined with chronic cardiovascular disease (e.g. congenital heart disease, congestive heart failure, or coronary artery disease, but doesnt include hypertension without any other cardio-related symptoms);
  4. Combined with hematological system diseases (e.g. chronic myelogenous leukemia, lymphocytic leukemia, myelodysplastic syndrome, aplastic anemia);
  5. Neurodevelopmental disorders, include cerebrum, spinal cord, Peripheral nerve and muscle disorders (e.g. cerebral palsy, epilepsy[epileptic seizure disorder], stroke, dysgnosia, Moderate to severe dysplasia, myodystrophy, or spinal cord injury);
  6. Poor control of chronic metabolic and endocrine diseases;
  7. Immunosuppression (long-term use of immunosuppressant, immunocom promise caused by infection by HIV or malignant tumour);
  8. Obese people[BMI>30, BMI=Weight(kg)/Height(m2)] 5.Long-term take aspirin under 19 years old; 6.White blood cell count>11.0×109/L, or the proportion of neutrophils >80%, or need systemic antibacterial therapy; 7.24 hours before the visit, the patients have received antiviral treatment for influenza; 8.The patients have received Influenza vaccine or research monoclonal antibody in a year; 9.ALT and AST is equal or greater than 1.5 times of upper limit of normal, Scr is greater than upper limit of normal; 10.Suspected or really have a history of alcohol or drug abuse; 11.Gestation (have a positive pregnancy test), lactating women, or have a family planning within the next 6 months; 12.The patients have participated in other clinical trials within 3 months; 13.The investigator considers it inappropriate to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
The time of fever relieving | day 3
  After the first dose, the time of subjects' armpit temperature reduced to 37.3℃, and no longer increases in 24h.

SECONDARY OUTCOMES:
symptom alleviating time of influenza | day 3 and day 5
  The area under the curve (AUC) of the decline in the subjects' influenza symptom total score.
Percentage of subjects with influenza complications Percentage of subjects with influenza complications | day 3 and day 5
  Percentage of subjects with influenza complications, e.g. be hospitalized, death, sinusitis, otitis media, bronchitis, pneumonia, and so on.
Percentage of antipyretic drugs used | day 3 and day 5
  Percentage of the subjects used paracetamol.
Percentage of virus positive to negative | day 3 and day 5
  Percentage of subjects' influenza virus positive change to negative

CONTACTS AND LOCATIONS:
Overall Officials: Qingquan Liu, Professor, Study Chair — Beijing Chinese Medicine Hospital affiliated to Capital Medical University

IPD SHARING:
Plan to Share IPD: No